CLINICAL TRIAL: NCT06087068
Title: A Prospective, Single-arm Phase II Study of Thyroxine Replacement Therapy After Lobectomy for Low-risk Papillary Thyroid Carcinoma
Brief Title: Thyroxine Replacement Therapy After Lobectomy for Low-risk Papillary Thyroid Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, liu jie, clinical professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cancer
Record Dates: First submitted 2023-10-08; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Cancer; Surgery; Recurrence
Keywords: thyroid cancer; lobectomy; TSH replacement; recurrence
MeSH Terms: conditions — Thyroid Neoplasms; Recurrence | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: The treatment goal after lobectomy was to control TSH within the normal reference range (0.4-5 mU/L)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test group (Experimental): The treatment goal after lobectomy was to control TSH within the normal reference range (0.4-5 mU/L)
  Interventions: Drug: Thyroxine

INTERVENTIONS:
Drug: Thyroxine — The treatment goal after lobectomy was to control TSH within the normal reference range (0.4-5 mU/L)

SUMMARY:
Papillary thyroid carcinoma (PTC) is the most common thyroid cancer and has a good prognosis.According to the 2015 American thyroid association (ATA) guidelines, no gross extrathyroidal extension and the number of pathological lymph node micrometastases (<0.2cm) ≤5 were defined as the low recurrence risk group. After total thyroidectomy and radioiodine treatment, the probability of disease-free status (irritant Tg<1ng/ml, no evidence of other disease recurrence) is about 78%-91%, and the probability of structural recurrence is about 1%-10%. In recent years, due to the further understanding of PTC, surgeons tend to become more conservative in treatment, such as active observation or reducing the extent of surgery. The indication for lobectomy has been extended to tumors <4cm without extrathyroidal extension and clinical lymph node metastasis. For patients treated with lobectomy, current guidelines recommend that Thyroid Stimulating Hormone (TSH) be controlled at 0.5-2 mU/L, but evidence on the prognostic benefits of this TSH inhibition range is lacking.In recent years, a number of studies have suggested that if postoperative TSH in low-risk patients after lobectomy is acceptable within the reference range, it means that a considerable number of patients have a high probability of not receiving thyroxine replacement therapy after surgery, which can significantly improve their quality of life.A previous retrospective study from our institute showed no significant association between TSH levels after lobectomy and prognosis.The aim of this study was to evaluate the benefits and risks of postoperative TSH levels within the reference range (0.4-5 mU/L) in patients with low-risk papillary thyroid cancer who underwent lobectomy.In order to improve the effect of longer recurrence and death time of PTC, the investigators also performed postoperative thyroglobulin and its antibody for short-term treatment response evaluation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18-70 years old, ECOG score 0-2;
* (2) Patients with the maximum diameter of unilateral thyroid nodules ≤4.0cm by ultrasound, papillary thyroid carcinoma diagnosed by preoperative cytology (Bethesda grade VI) or intraoperative freezing, and planned to undergo thyroid lobectomy;
* (3) No clinical lymph node metastasis (cN0);No extrathyroidal extension, and the number of pathological lymph node micrometastasis (<0.2cm) was ≤5.
* (4) no serious medical diseases and major organ dysfunction, such as blood routine, liver, kidney, heart, lung function; No previous history of other head and neck malignancies, no history of neck radiation, no history of deep neck surgery (skin mass excision except clinical);
* (5) Fully understand this study, have the ability to complete treatment, have follow-up conditions and voluntarily sign informed consent.

Exclusion Criteria:

* (1) History of malignancy in other sites (previous or simultaneous), excluding curable non-melanoma skin cancer and cervical carcinoma in situ;
* (2) The contralateral thyroid nodules were evaluated by preoperative ultrasound, and the patients with suspicious nodules who underwent fine-needle aspiration cytology and could not confirm the benign or malignant nodules (Bethesda grade I, III-V) were excluded.
* (3) Cervical lymph node metastasis was evaluated before surgery. Cytological aspiration and Tg eluent determination were performed on suspicious lymph nodes. If cytology was negative and Tg eluent was not higher than the normal range, it was not considered as exclusion criteria. The patients who were sent for intraoperative examination and showed metastasis were excluded.
* (4) cytological aspiration or intraoperative freezing suspected non-papillary thyroid carcinoma (follicular carcinoma, medullary carcinoma, poorly differentiated or undifferentiated carcinoma) or high-risk subtypes of papillary thyroid carcinoma (high cell type);
* (5) pregnant or lactating women；
* (6) A history of drug use or drug abuse within the past 1 year;
* (7) Participants who had participated in other clinical trials within 4 weeks before enrollment;
* (8) The patient is unable to accept the preservation of the contralateral gland or cannot cooperate with subsequent thyroid hormone replacement therapy.
* (9) The investigator assesses subjects who are unsuitable for the trial for other reasons, or who are not expected to complete the study.

Ages: 18 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence | 2 year
  recurrence-free survival

SECONDARY OUTCOMES:
thyroid function | 1 year; 2 year
  biochemical incomplete (rising serum Tg)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China